CLINICAL TRIAL: NCT05694455
Title: Clinical Utility of Longitudinal Measurement of Hemodynamic Incoherence and Endothelial
Brief Title: Micro and Macro Circulation in Sepsis
Acronym: DAISY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Ivor Douglas, Chief Pulmonary Critical Care, Denver Health and Hospital Authority
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 22-0349
Record Dates: First submitted 2023-01-05; First posted 2023-01-23 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Sepsis; Septic Shock
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Urine Specimen Collection

STUDY DESIGN:
Intervention Model Description: Patients diagnosed with septic shock in the emergency department admitted to the hospital will be enrolled within 4 hours of the emergency physician's decision to admit the patient to the hospital.
  On enrollment, On enrollment and at hours 10-14, 22-26, and 44-48, the research team will assess micro hemodynamic incoherence and Macro hemodynamic incoherence as well as the total amount of IV fluids and vasoactive medications administered, demographics, Charlson morbidity scale and Sofa score.
  Healthy controls will have sublingual microscopy and urine collection performed at time of intubation for elective procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Septic Patient Interventions (Other): Septic Patients will have all interventions performed: Urine collection, Passive Leg Raise, Ultrasound and sublingual microscopy
  Interventions: Diagnostic Test: Starling Stroke Volume (Starling SV)- Passive Leg Raise; Diagnostic Test: Microscan Sublingual Microscopy; Diagnostic Test: Venous Excess Ultrasound Scoring (VExUS); Other: Urine Collection
- Control Patient Interventions (Other): Control patients will have urine collection and sublingual microscopy performed when intubated
  Interventions: Diagnostic Test: Starling Stroke Volume (Starling SV)- Passive Leg Raise; Other: Urine Collection

INTERVENTIONS:
Diagnostic Test: Starling Stroke Volume (Starling SV)- Passive Leg Raise — All septic patients will have a passive leg raise performed with the assistance of an Starling SV device to look at Stroke Volume change. This will be performed at admission and 4 hours after admission. This intervention will not be performed on healthy controls
  Other Names: Baxter Starling Stroke Volume (SV)
Diagnostic Test: Microscan Sublingual Microscopy — All septic patients will have sublingual microscopic images performed at admission, 8-16 hours, 48 hours and 72 hours. Control patients will have a sublingual microscope imaging performed after intubation for the elective procedure. This is a process of a 2cm probe tip gently placed on patients' mouth and 3 different images of 5-8 seconds are recorded.
  Other Names: Microvision Sublingual Microscopy
  Arms: Septic Patient Interventions
Diagnostic Test: Venous Excess Ultrasound Scoring (VExUS) — All septic Patients will have this performed on all patients at admission, 8-16 hours, 48 hours and 72 hours. Ultrasound images and blood flow waves will be collected of the Inferior Vena Cava diameter, hepatic vein, portal vein, renal veins and scored using the Venous Excess Ultrasound (VExUS scale). Healthy controls will not have ultrasound performed
  Arms: Septic Patient Interventions
Other: Urine Collection — The urine assay is collected passively from the patient will be ran through a Dimethylmethylene blue (DMMB assay)- could provide future beneficial information to resuscitation efforts. This will be performed on all septic patients at admission, 8-16 hours, 48 hours and 72 hours. Urine will be collected on healthy controls at time of intubation for elective procedure.

SUMMARY:
Purpose: To assess the prognostic role of Handheld Vital Microscopy (HVM) and evaluate levels of endothelial glycocalyx (eGC) breakdown in patients demonstrating Hemodynamic Incoherence (HI), to elucidate a mechanistic link between the eGC and HI in order to inform prognostic enrichment of future resuscitation trials. We will serially evaluate microhemodynamics (MiH) and macro hemodynamics (maH) and the perfused boundary region (PBR, an visual proxy for eGC thickness) using HVM, and a validated circulating biomarker of eGC integrity.

DETAILED DESCRIPTION:
There are few reliable prognostic indicators in early sepsis to predict disease progression, in part because the pathophysiologic mechanism of vascular dysregulation remains incompletely understood. The global Coronavirus Disease 2019 (COVID-19) pandemic has increased the number of patients with sepsis, straining hospital systems and illustrating the need for research into prognostic and therapeutic strategies. An important area of research is the role of the eGC, a thin vascular lining composed of proteoglycans, glycosaminoglycan side-chains, and plasma proteins that play a central role in microvascular homeostasis, the function of which is compromised in sepsis. Another growing field of inquiry is the phenomenon of HI, a condition in which MiH remain dysfunctional despite normalization of conventionally targeted MaH measures such as mean arterial pressure (MAP), leading to poor end-organ perfusion. It has been hypothesized that HI due to persistently deranged MiH and reduced end-organ perfusion result in an ongoing state of "microvascular shock", leading to worsening end-organ damage despite apparent normalization of conventionally targeted parameters. Importantly, HI has been shown to predict poor patient outcomes, with abnormal MiH predicting patient mortality despite normalization of MAP after administration of vasoactive medications. MiH measures have also been shown to differ significantly between septic patients and healthy controls. In one study of a large sepsis cohort, MiH parameters were predictive of adverse outcomes, while MaH parameters were not, suggesting that MiH measurements, and HI in particular may be more sensitive than conventional measures for predicting outcomes in sepsis. One hypothesis is that HI in sepsis is mediated by degradation of the eGC, with subsequent loss of microvascular homeostasis, though the role of the eGC as a vascular barrier remains controversial.

One question that remains is whether or not microvascular changes can predict patient outcomes in patients judged to be adequately fluid resuscitated, as measured by MAP or Starling Stroke Volume/Non-invasive cardiac monitor (NICOM) testing.

ELIGIBILITY:
Inclusion Criteria:

Septic Patient Cohort:

1. Greater than or equal to 18 years of age
2. Diagnosed with sepsis or septic shock
3. Require admission to the Hospital

Control Cohort:

1. Greater than or equal to 18 years of age
2. Undergoing elective surgery requiring intubation and general anesthesia

Exclusion Criteria:

Patients with any of the following characteristics will be excluded

1. Less than 18 years old
2. Chronic Kidney disease on dialysis
3. Currently pregnant
4. Incarcerated persons

Control Cohort:

1. Less than 18 years old
2. History of Chronic Kidney disease on dialysis, uncontrolled diabetes, cirrhosis, heart failure, or nephritic or nephrotic syndromes.
3. Currently pregnant
4. Incarcerated persons

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Initiation and Duration Renal Replacement Therapy | 90 day
  Renal Replacement Therapy will be monitored while hospitalized for Sepsis/Septic Shock for initiation and days receiving Renal replacement will be counted.

SECONDARY OUTCOMES:
Rate of Inpatient Mortality | 90 day
  Patient Death while hospitalized for the admission of Sepsis/Septic Shock
Rate of 90 day survival | 90 day
  Patient death within 90 days of admission to the hospital for Sepsis/Septic Shock

CONTACTS AND LOCATIONS:
Locations (1):
- Denver Health Medical Center, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
currently individual participant data will not be made available to other researchers